CLINICAL TRIAL: NCT02215356
Title: Icotinib With Concurrent Radiotherapy Versus Etoposide/Cisplatin With Concurrent Radiotherapy in Stage III Non-small Cell Lung Cancer With EGFR 19/21 Mutation
Brief Title: Icotinib With Concurrent Radiotherapy Versus Chemotherapy With Concurrent Radiotherapy in Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV66
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Chemoradiotherapy; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoradiotherapy (Active Comparator): Etoposide 50mg/m2, ivgtt, d1-d5, cisplatin 50mg/m2, ivgtt, d1 and d8, every 28 days for a cycle, a total of 2 cycles, while chest radiotherapy (total dose 60-66Gy, 2Gy per time, once a day, five times a week, a total of 30-33 times). Progressive patients will be administered oral icotinib 125 mg three times daily.
  Interventions: Drug: Chemoradiotherapy
- Icotinib with concurrent radiotherapy (Experimental): Chest radiotherapy (total dose 60-66Gy, 2Gy per time, once a day, five times a week, a total of 30-33 times), while icotinib 125mg three times daily (375 mg per day) by mouth. Maintenance icotinib will be administered after radiotherapy. Progressive patients will receive chemotherapy, using the platinum-based two-drug chemotherapy regimen.
  Interventions: Drug: Icotinib with concurrent radiotherapy

INTERVENTIONS:
Drug: Icotinib with concurrent radiotherapy — Icotinib: 125 mg is administered orally three times per day.
  Other Names: Icotinib; Comana; BPI-2009
  Arms: Icotinib with concurrent radiotherapy
Drug: Chemoradiotherapy — Etoposide 50mg/m2, ivgtt, d1-d5; cisplatin 50mg/m2, ivgtt, d1 and d8, every 28 days for a cycle, a total of 2 cycles
  Other Names: VP16; DDP
  Arms: Chemoradiotherapy

SUMMARY:
This randomised, multi-center, controlled trial is designed to assess the efficacy and safety of icotinib with concurrent radiotherapy versus chemotherapy with concurrent radiotherapy in non-small cell lung cancer

DETAILED DESCRIPTION:
This randomised, multi-center, controlled trial is designed to assess the efficacy and safety of icotinib with concurrent radiotherapy versus etoposide/cisplatin with concurrent radiotherapy in stage III non-small cell lung cancer with EGFR 19/21 Mutation, the primary endpoint is progression-free survival

ELIGIBILITY:
Inclusion Criteria:

* Unresectable stage IIIA / IIIB non-small cell lung cancer with EGFR 19/21 mutation
* No previous systemic anticancer therapy
* Measurable lesion according to RECIST with at least one measurable lesion not previously irradiated, unless disease progression has been documented at that site
* ECOG Performance Status of 0 to 1

Exclusion Criteria:

* Prior treatment with anti-EGFR (the epidermal growth factor receptor) monoclonal antibody or small molecular compounds therapy such as gefitinib, erlotinib or cetuximab
* Evidence of clinically active Interstitial Lung Diseases (patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded)
* Known severe hypersensitivity to icotinib or any of the excipients of this product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months

SECONDARY OUTCOMES:
Overall survival | 36 months
Objective response rate | 8 weeks
Adverse events | 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Lvhua Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Xiaolong Fu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (26):
- China (26):
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - People's Liberation Army 307 Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Union Medical College Hospital, Beijing, Beijing Municipality
  - Dongguan City People's Hospital, Dongguan, Guangdong
  - Sun Yat-sen Cancer Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Hunan Provincial Tumor Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - Tumor Hospital of Jilin Province, Changchun, Jilin
  - Liaoning Provincial Tumor Hospital, Shenyang, Liaoning
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanxi Tumor Hospital, Taiyuan, Shanxi
  - Sichuan Provincial Tumor Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Tumor Hospital of Yunnan Province, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang